CLINICAL TRIAL: NCT04345419
Title: Remdesivir in COVID-19 Treatment: A Randomised Trial
Brief Title: Remdesivir Efficacy in Coronavirus Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, assistant professor of tropical medicine and infectious diseases, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID 19 treatment
Record Dates: First submitted 2020-04-11; First posted 2020-04-14 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: COVID
MeSH Terms: interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remdesivir (Experimental): Remdesivir with standard of care treatment standard of care treatment
  Interventions: Drug: Remdesivir; Other: Standard of care treatment
- Standard of care (Placebo Comparator): Standard of care treatment alone.
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Drug: Remdesivir — Remdesivir as antiviral drug
  Arms: Remdesivir
Other: Standard of care treatment — Standard of care treatment

SUMMARY:
COVID 19 treatment using Remedesvir.

DETAILED DESCRIPTION:
COVID 19 treatment using Remedesvir. Is this drug effective?

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 patients

Exclusion Criteria:

* allergy or contraindication to the drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with improvement or mortality | 6 months
  the estimated number of patients with improvement or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, ass. prof., Principal Investigator — Tanta University Faculty of medicine
Locations (1):
- Tanta university hospital, Assuit University, Ainshams University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483